CLINICAL TRIAL: NCT07122284
Title: Characterization of Gut Microbiota and Metabolic Profiles in Patients With Helicobacter Pylori Infection and Small Intestinal Bacterial Overgrowth Based on Metagenomic and Metabolomic Analyses
Brief Title: Gut Microbiome-Metabolome Profiling in H. Pylori-SIBO Comorbidity
Status: Completed | Type: Observational
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Principal Investigator, Yucheng Zhu, Deputy Chief Physician, Zhongshan Hospital (Xiamen), Fudan University
Other Study IDs: ZYC-SIBO2025
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Gut Microbiota; Metabolic Profiles; Helicobacter Pylori Infection; Small Intestinal Bacterial Overgrowth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Metagenomics and metabolomics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: H. pylori-positive and SIBO-positive group
  Interventions: Diagnostic Test: 13C-Urea Breath Test; Diagnostic Test: Hydrogen-Methane Breath Test
- Group B: H. pylori-negative and SIBO-positive group
  Interventions: Diagnostic Test: 13C-Urea Breath Test; Diagnostic Test: Hydrogen-Methane Breath Test
- Group C: H. pylori-positive and SIBO-negative group
  Interventions: Diagnostic Test: 13C-Urea Breath Test; Diagnostic Test: Hydrogen-Methane Breath Test
- Group D: H. pylori-negative and SIBO-negative group
  Interventions: Diagnostic Test: 13C-Urea Breath Test; Diagnostic Test: Hydrogen-Methane Breath Test

INTERVENTIONS:
Diagnostic Test: 13C-Urea Breath Test — Participants underwent the 13C-urea breath test following a standardized protocol to detect active Helicobacter pylori (H. pylori) infection. After an overnight fast (≥8 hours), baseline breath samples were collected by exhaling gently through a straw. Participants then ingested 75 mg of 13C-labeled urea dissolved in 50 mL of citric acid solution to delay gastric emptying and maximize urease exposure. A second breath sample was collected 30 minutes post-ingestion using identical procedures.
Diagnostic Test: Hydrogen-Methane Breath Test — Participants underwent a standardized hydrogen-methane breath test to evaluate for small intestinal bacterial overgrowth (SIBO) or carbohydrate malabsorption. After a 12-hour overnight fast, baseline breath samples were collected via controlled end-expiratory exhalation. Participants then ingested a substrate solution.

SUMMARY:
Patients with concurrent Helicobacter pylori infection and small intestinal bacterial overgrowth (SIBO) represent a clinically challenging subgroup, often experiencing refractory gastrointestinal symptoms and diminished treatment responses. Current evidence indicates that individuals infected with H. pylori may related SIBO as a comorbidity; however, the synergistic effects of these conditions on gut ecosystem homeostasis remain poorly understood. To address this knowledge gap, we employed a dual-omics approach that combined shotgun metagenomic sequencing with liquid chromatography-mass spectrometry (LC-MS) metabolomic profiling. This methodology allowed for a comprehensive mapping of microbial community structures, including species-level taxonomy and functional pathways, as well as host-microbiota co-metabolism signatures in fecal samples.

DETAILED DESCRIPTION:
Patients presenting with concurrent Helicobacter pylori infection and small intestinal bacterial overgrowth (SIBO) constitute a clinically challenging subgroup characterized by refractory gastrointestinal symptoms and diminished responses to standard therapeutic interventions. Current evidence supports an association between H. pylori infection and an increased prevalence of SIBO as a comorbidity. However, the synergistic effects of these two conditions on the fundamental mechanisms governing gut ecosystem homeostasis - particularly concerning microbial community dynamics, functional metabolic output, and host-microbial interactions - remain poorly understood, representing a significant knowledge gap.

To systematically address this gap and elucidate the complex interplay, we implemented an integrated dual-omics analytical approach. This methodology combined shotgun metagenomic sequencing of fecal samples with liquid chromatography-mass spectrometry (LC-MS) metabolomic profiling. This powerful combination enables a comprehensive mapping of the gut ecosystem by simultaneously characterizing: Host-Microbiota Co-Metabolism Signatures: Revealing the metabolic landscape through the detection and quantification of metabolites derived from microbial activity, host metabolism, and crucially, their interactions (co-metabolism) within the fecal metabolome.

This multimodal strategy offers an unprecedented, holistic view of the perturbations induced by the co-occurrence of H. pylori infection and SIBO, moving beyond singular aspects to capture the integrated functional and compositional state of the gut ecosystem.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years;
* All enrolled patients underwent both the 13C-urea breath test (13C-UBT) and hydrogen-methane breath test (HMBT).

Exclusion Criteria:

* Coexistence of significant concomitant illnesses, including heart disease, renal failure, hepatic disease, previous abdominal surgery, lactation, or pregnancy;
* Patients who had used probiotics and antibiotics in the past 12 weeks;
* Unwillingness to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational cohort of adult patients (aged 18-65 years) with concomitant Helicobacter pylori infection and small intestinal bacterial overgrowth (SIBO) was enrolled at Zhongshan Hospital (Xiamen), Fudan University.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
13C-Urea Breath Test | day 0, Patient baseline levels at enrollment
  The 13C-Urea Breath Test (13C-UBT) is a non-invasive, highly specific diagnostic assay used to detect active Helicobacter pylori (H. pylori) infection in the gastric mucosa. It leverages the bacterium's unique enzymatic activity-urease production-to metabolize ingested labeled urea, resulting in measurable changes in exhaled breath CO₂ isotopic composition.
Hydrogen-Methane Breath Test | day 0, Patient baseline levels at enrollment
  The Hydrogen-Methane Breath Test (HMBT) is a non-invasive, gold-standard diagnostic tool for detecting small intestinal bacterial overgrowth (SIBO) and carbohydrate malabsorption disorders . It quantifies microbial fermentation activity in the gut by measuring gaseous metabolic end-products (H₂ and CH₄) in exhaled breath following substrate administration.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, M.D., Study Director — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Zhongshan Hospital (Xiamen), Fudan University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Zhu D, Li S, Dai Y, Teng G, Wang W. Influence of Helicobacter pylori Infection and Eradication on Small Intestinal Bacterial Overgrowth and Abdominal Symptoms. Dig Dis Sci. 2024 Apr;69(4):1293-1301. doi: 10.1007/s10620-024-08279-y. Epub 2024 Feb 15. PMID 38363519
- [Result] Nelson JM, Rizzo JM, Greene RK, Fahlstrom K, Troost JP, Helfrich YR, Nakamura M. Evaluation of Helicobacter pylori and Small Intestinal Bacterial Overgrowth in Subjects With Rosacea. Cureus. 2024 Oct 25;16(10):e72363. doi: 10.7759/cureus.72363. eCollection 2024 Oct. PMID 39583431